CLINICAL TRIAL: NCT04323137
Title: Encouraging Flu Vaccination Among High-Risk Patients Identified by a Machine-Learning Model of Flu Complication Risk
Brief Title: Encouraging Flu Vaccination Among High-Risk Patients Identified by ML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christopher F Chabris, PhD, Faculty Co-Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-0290; 5P30AG034532-12 (NIH)
Record Dates: First submitted 2020-03-19; First posted 2020-03-26 (Actual); Results first posted 2022-11-07 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Influenza; Vaccination; Health Promotion; Health Behavior; Risk Reduction
Keywords: Flu Vaccine; Choice Architecture; Machine Learning; Perceived Credibility
MeSH Terms: conditions — Influenza, Human; Health Behavior; Risk Reduction Behavior | interventions — Numbers Needed To Treat

STUDY DESIGN:
Intervention Model Description: Patients from the high-risk sample will be randomly assigned to one of 4 groups:
  1. Control: group that receives no additional pro-vaccination intervention beyond Geisinger's normal efforts.
  2. High Risk Only: group that receives messages telling them they have been identified to be at high risk for flu complications without specifying how/why Geisinger believes this to be the case
  3. High Risk Based on Medical Records: group that receives messages telling them they have been identified to be at high risk for flu complications via analysis of their medical records
  4. High Risk Based on Algorithm: group that receives messages telling them they have been identified to be at high risk for flu complications via analysis of their medical records by AI/ML
     Two additional groups will be monitored for outcome data:
  5. Sub-threshold patients: patients who are in the top 11-20% of risk
  6. Household members: patients who share an address with target patients
Who Masked: Participant, Care Provider
Masking Description: Participants (i.e., patients) will not be informed specifically of their assignment to different arms throughout the study. Providers who prescribe vaccination and diagnose conditions will not be randomized to study arms or informed of patient assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (No Intervention): This group receives no additional pro-vaccination intervention beyond the health system's normal efforts. Although some patients are currently targeted for flu vaccination encouragement due to a non-ML assessment that they are at high risk for complications, these patients are not told that they are at high risk or that they have been targeted.
- High risk only (Experimental): This group receives messages telling them they have been identified to be at high risk for flu complications without specifying how or why the health system believes this to be the case.
  Interventions: Behavioral: Risk reduction
- High risk based on medical records (Experimental): This group receives messages telling them they have been identified to be at high risk for flu complications via analysis of their medical records.
  Interventions: Behavioral: Risk reduction; Behavioral: Medical records-based recommendation
- High risk based on algorithm (Experimental): This group receives messages telling them they have been identified to be at high risk for flu complications via analysis of their medical records by an AI/ML system.
  Interventions: Behavioral: Risk reduction; Behavioral: Medical records-based recommendation; Behavioral: Algorithm-based recommendation
- Sub-threshold patients (No Intervention): Patients in this group is in the top 11-20% of risk for flu and complications, slightly lower risk than those included in the intervention, who are in the top 10% of risk for flu and complications. This group of patients does not receive an intervention, but are monitored for flu shots as a comparison to target patients.
- Household members (No Intervention): This group of patients share an address with target high-risk patients (in arms 1-4). This group does not receive an intervention but is monitored for spillover effects of the intervention.

INTERVENTIONS:
Behavioral: Risk reduction — Mailed letter, SMS, and/or patient portal message
  Arms: High risk based on algorithm; High risk based on medical records; High risk only
Behavioral: Medical records-based recommendation — Mailed letter, SMS, and/or patient portal message
  Other Names: Credibility
  Arms: High risk based on algorithm; High risk based on medical records
Behavioral: Algorithm-based recommendation — Mailed letter, SMS, and/or patient portal message
  Other Names: Credibility
  Arms: High risk based on algorithm

SUMMARY:
The purpose of the current study is to test different interventions to determine the most effective way to promote flu vaccine uptake in a high-risk population identified by an "artificial intelligence" (AI) or machine learning (ML) algorithm. The specific aims are:

1. Evaluate the effect on flu vaccination rates of informing health-system patients who are identified by an ML analysis of EHR data to be at high risk for flu complications that they are at high risk with either (a) no additional explanation, (b) an explanation that this determination comes from an analysis of their medical records, and (c) the additional explanation that an AI or ML algorithm made this determination.
2. Evaluate the effects of the same three interventions on diagnoses of flu in the same patients.

DETAILED DESCRIPTION:
Background

On average, 8% of the US population gets sick from flu each flu season (Tokars et al. 2018). Since 2010, the annual disease burden of influenza has included 9-45 million illnesses, 140,000-810,000 hospitalizations, and 12,000-61,000 deaths (CDC 2020). The CDC recommends the flu vaccination to everyone aged 6+ months, with rare exception; almost anyone can benefit from the vaccine, which can reduce illnesses, missed work, hospitalizations, and death (CDC 2019a). Flu vaccination will be especially important for high-risk patients during the COVID-19 pandemic so that flu cases are reduced and resources conserved.

While most recover from influenza without treatment, the elderly, those with comorbidities, and other high-risk individuals can experience complications such as pneumonia, other respiratory illness, and death. Geisinger, a large health system in Pennsylvania and New Jersey, has partnered with Medial EarlySign (Medial; www.earlysign.com) to develop a machine learning (ML) algorithm to identify patients at risk for serious (moderate to severe) flu-associated complications on the basis of their existing electronic health record (EHR) data. Geisinger will deploy this system during the 2020-21 flu season and contact the identified patients with special messages (in addition to standard efforts made by the health system every flu season) to encourage vaccination. Flu vaccination will be especially important for high-risk patients during the COVID-19 pandemic so that flu cases are reduced and resources conserved.

Published results suggest Medial's ML systems identify high-risk patients in other contexts (Goshen et al., 2018; Zack et al., 2019). However, there is little evidence about (a) whether informing patients they are at high risk makes them more likely to receive vaccination; (b) how patients react to being told their risk status is the result of an analysis of their health records; and (c) whether informing patients their risk status has been determined by an "algorithm," by "machine learning," and/or by "artificial intelligence" will increase or decrease their likelihood of getting vaccinated. This study will address these gaps in the literature, which are especially important in light of the anticipated future growth of AI/ML system use throughout healthcare.

Medial's algorithm is an example of how interoperable health information exchange (HIE)-the ability for health information technology to share patient data-can improve the efficiency and effectiveness of healthcare. However, patients may not appreciate these benefits or the fact that healthcare has become substantially more integrated and collaborative. A systematic review of patient privacy concerns about HIE found that 15-74% of patients expressed privacy concerns, depending on the study, and concluded that patient perspectives remain poorly understood. A flu outreach message that explicitly references a review of patient medical records might backfire as patients react badly to a sense they have lost control of their health records.

There is conflicting evidence on how people respond to advice or information that comes from an algorithm or machine. Dietvorst et al. (2015) documented a pattern of "algorithm aversion," in which people choose inferior human over superior algorithmic forecasts, especially after they observed the algorithm make an error. In contrast, Logg et al. (2018) described "algorithm appreciation," in which people followed advice more when they thought it came from algorithms than when they thought it came from human beings. Finally, Bigman and Gray (2019) found aversion to algorithms that make "moral decisions," including a (fictitious) medical decision of choosing whether or not to operate on a high-risk patient. In the current setting, the algorithm is merely advising patients on taking an action (an annual flu shot) that is already the standard of care, and there is no opportunity to observe an erroneous recommendation, so the hypothesis is that "algorithm appreciation" will cause people to react positively to being informed of the algorithm's role. Thus, this study will address two important research questions:

1. Does informing patients that they are at high risk for flu complications (a) increase the likelihood that they will receive flu vaccine; and (b) decrease the likelihood that they receive diagnoses of flu and/or flu-like symptoms in the ensuing flu season?
2. Does informing patients that their high-risk status was determined (a) by analyzing their medical records (vs. by no specified method); and (b) by an AI/ML algorithm* analyzing their medical records (as opposed to via unspecified methods or human medical records analysis) affect the likelihood that they receive the flu vaccine and/or diagnoses of flu and/or flu-like symptoms in the ensuing flu season?

Our specific aims are:

1. Evaluate the effect on flu vaccination rates of informing health-system patients who are identified by an ML analysis of EHR data to be at high-risk for flu complications that they are at high risk with either (a) no additional explanation, (b) an explanation that this determination comes from an analysis of their medical records, and (c) the additional explanation that an AI or ML algorithm made this determination.
2. Evaluate the effects of the same three interventions on diagnoses of flu in the same patients.

Research Strategy

Included in the study will be current Geisinger patients 17+ years of age with one or more visits to a Geisinger primary care physician (PCP) between January 1, 2008 and January 30, 2020 and no contraindications for flu vaccine. Medial will provide flu-complication risk scores from their ML algorithm (based on coded EHR data), on the basis of which the top 10% of patients at highest risk will be included. Based on prior behavior and other predictors in a second ML model, Medial will also provide the likelihood each patient will get vaccinated during the study flu season; these values and the primary risk scores will be used as covariates in exploratory data analyses. The anticipated number of patients in the top 10% of risk is 56,000.

On average in the last 3 flu seasons, 55% of Geisinger patients aged 65+ are vaccinated each season, so we will use this as a proxy base rate for a control condition in our power analysis. The study will have 92% power to detect a 2% absolute difference or greater in the vaccination outcome between conditions (55% vs 57%, two-tailed alpha of .05), on the assumption that each condition will have 56,000/4=14,000 patients. For the rarer outcome of flu diagnosis, we have 95% power to detect a 0.8% absolute difference or greater-from an estimated 3.9% rate in this high-risk population (based on the CDC estimate for people age 65+ [Tokars et al., 2018]) to a 3.1% rate.

The primary study outcomes will be the rates of flu vaccination and flu diagnoses during the 2020-21 season (September-March) by targeted patients. Secondary, exploratory outcomes will also be measured: Rates of flu vaccination and diagnoses by fellow household members of targeted patients; rates of flu vaccination and diagnoses by non-targeted patients who were assigned a risk score that fell just below the cutoff of targeted patients ("sub-threshold risk"); rates of flu complications and flu-like symptoms among targeted patients, household members, and those at sub-threshold risk; and rates of other relevant healthcare utilization outcomes such as ER visits and hospitalizations.

Generalized linear mixed models (GLMMs) will examine the primary study outcomes as a function of the study arms (between-subjects), with patient-visited PCPs and/or clinics included as random effects variables, assuming high intraclass correlation coefficients. GLMMs will specify a binary distribution and log-link function in the case of dichotomous outcome variables (e.g., flu vaccination, flu diagnosis), and a negative binomial distribution and log-link function in the case of any highly positively skewed count variables such as ER visits and hospitalizations (where over-dispersion typically remains in the case of a Poisson distribution model). For these exploratory analyses, within-patient change (from the same period one year earlier) will also be analyzed. Also, each patient will receive the same type of communication (a/b/c/d) via up to three modalities-printed letter to their mailing address, SMS to their mobile phone, and/or secure message via Geisinger's patient portal-depending on what information is on file for each patient. The communication channels used for each patient will be covariates in later analyses.

*Note: The study will not necessarily use the terms "AI," "ML," or "algorithm" in the messages to groups b, c, and d; instead, these messages will be designed to be readable and comprehensible by the patient audience while still including the key concepts that differentiate the interventions from one another.

ELIGIBILITY:
Inclusion Criteria:

* Current Geisinger patient at the time of study
* Falls in the top 10% of patients at highest risk, as identified by the flu-complication risk scores of Medial's machine learning algorithm (which operates on coded EHR data)
* May limit inclusion to patients that are under Geisinger primary care, depending on algorithm performance of patients who have non-Geisinger PCPs

Exclusion Criteria:

* Has contraindications for flu vaccination
* Has opted out of receiving communications from Geisinger via all of the modalities being tested

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117649 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chabris, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data and code are available in the OSF repository at the url below in the folder ClinicalTrials.gov data/Study 1.
URL: https://osf.io/mqbux/

REFERENCES:
- [Background] Bigman YE, Gray K. People are averse to machines making moral decisions. Cognition. 2018 Dec;181:21-34. doi: 10.1016/j.cognition.2018.08.003. Epub 2018 Aug 11. PMID 30107256
- [Background] Dietvorst BJ, Simmons JP, Massey C. Algorithm aversion: people erroneously avoid algorithms after seeing them err. J Exp Psychol Gen. 2015 Feb;144(1):114-26. doi: 10.1037/xge0000033. Epub 2014 Nov 17. PMID 25401381
- [Background] Goshen R, Choman E, Ran A, Muller E, Kariv R, Chodick G, Ash N, Narod S, Shalev V. Computer-Assisted Flagging of Individuals at High Risk of Colorectal Cancer in a Large Health Maintenance Organization Using the ColonFlag Test. JCO Clin Cancer Inform. 2018 Dec;2:1-8. doi: 10.1200/CCI.17.00130. PMID 30652563
- [Background] Logg, J.M., Minson, J.A., & Moore, D.A. (2019). Algorithm appreciation: People prefer algorithmic to human judgment. Organizational Behavior and Human Decision Processes, 151, 90-103. https://doi.org/10.1016/j.obhdp.2018.12.005
- [Background] Shen N, Bernier T, Sequeira L, Strauss J, Silver MP, Carter-Langford A, Wiljer D. Understanding the patient privacy perspective on health information exchange: A systematic review. Int J Med Inform. 2019 May;125:1-12. doi: 10.1016/j.ijmedinf.2019.01.014. Epub 2019 Feb 1. PMID 30914173
- [Background] Rothberg MB, Haessler SD. Complications of seasonal and pandemic influenza. Crit Care Med. 2010 Apr;38(4 Suppl):e91-7. doi: 10.1097/CCM.0b013e3181c92eeb. PMID 19935413
- [Background] Tokars JI, Olsen SJ, Reed C. Seasonal Incidence of Symptomatic Influenza in the United States. Clin Infect Dis. 2018 May 2;66(10):1511-1518. doi: 10.1093/cid/cix1060. PMID 29206909
- [Background] Turner D, Wailoo A, Nicholson K, Cooper N, Sutton A, Abrams K. Systematic review and economic decision modelling for the prevention and treatment of influenza A and B. Health Technol Assess. 2003;7(35):iii-iv, xi-xiii, 1-170. doi: 10.3310/hta7350. PMID 14609480
- [Background] WHO Guidelines for Pharmacological Management of Pandemic Influenza A(H1N1) 2009 and Other Influenza Viruses. Geneva: World Health Organization; 2010 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK138515/ PMID 23741777
- [Background] Zack CJ, Senecal C, Kinar Y, Metzger Y, Bar-Sinai Y, Widmer RJ, Lennon R, Singh M, Bell MR, Lerman A, Gulati R. Leveraging Machine Learning Techniques to Forecast Patient Prognosis After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2019 Jul 22;12(14):1304-1311. doi: 10.1016/j.jcin.2019.02.035. Epub 2019 Jun 26. PMID 31255564
- [Background] Centers for Disease Control and Prevention. (2020). Disease Burden of Influenza. https://www.cdc.gov/flu/ about/burden/index.html (Jan 10).
- [Background] Centers for Disease Control and Prevention. (2019a). Who Needs a Flu Vaccine and When. https://www.cdc.gov/flu/prevent/vaccinations.htm (Oct 11).
- [Background] Centers for Disease Control and Prevention. (2019b). Flu Vaccination Coverage, United States, 2018-19 Influenza Season. https://www.cdc .gov/flu/fluvaxview/coverage-1819estimates.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Sub-threshold Patients: Patients in this group are in the top 11-20% of risk for flu and complications, slightly lower risk than those included in the intervention, who are in the top 10% of risk for flu and complications. This group of patients does not receive an intervention, but is monitored for flu shots as a comparison to target patients.
- Household Members: This group of patients share an address with target high-risk patients (in arms 1-4). This group does not receive an intervention but is monitored for spillover effects of the intervention.
  Note that some household members of target patients were also sub-threshold risk. Additionally, some of these patients were household members of more than one target patient.
  The numbers reported here reflect unique household members who were not also sub-threshold risk patients.
Period: Overall Study
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm | Sub-threshold Patients | Household Members
Started | 11667 | 11639 | 11652 | 11644 | 46898 | 24149
Completed | 11667 | 11639 | 11652 | 11644 | 46898 | 24149
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is the number of participants who were randomized to each arm. Some randomized participants were excluded from analysis if they were vaccinated prior to the study start date or if they were contraindicated for flu vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm | Sub-threshold Patients | Household Members | Total
Number analyzed (Participants) | 11667 | 11639 | 11652 | 11644 | 46898 | 24149 | 117649
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (19.3) | 57.9 (19.3) | 57.9 (19.2) | 57.6 (19.4) | 55.7 (19.5) | 47.1 (20) | 54.8 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7535 | 7514 | 7533 | 7438 | 29226 | 10744 | 69990
  Male | 4132 | 4125 | 4119 | 4206 | 17672 | 13405 | 47659
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 402 | 457 | 395 | 413 | 1684 | 1113 | 4464
  Not Hispanic or Latino | 11253 | 11159 | 11240 | 11207 | 45120 | 22777 | 112756
  Unknown or Not Reported | 12 | 23 | 17 | 24 | 94 | 259 | 429
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 22 | 21 | 15 | 22 | 47 | 32 | 159
  Asian | 32 | 37 | 28 | 31 | 189 | 124 | 441
  Native Hawaiian or Other Pacific Islander | 18 | 26 | 20 | 26 | 126 | 129 | 345
  Black or African American | 362 | 382 | 389 | 416 | 1603 | 1116 | 4268
  White | 11223 | 11159 | 11194 | 11136 | 44859 | 22674 | 112245
  Unknown or Not Reported | 10 | 14 | 6 | 13 | 74 | 72 | 189
Region of Enrollment [Number; unit: participants]
  United States | 11667 | 11639 | 11652 | 11644 | 46898 | 24149 | 44602

OUTCOME MEASURES:

1. Primary Outcome: Flu Vaccination Rate
Description: Patient received a flu vaccination
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: Participants were excluded from analysis if they were vaccinated prior to the study start date or if they were contraindicated for flu vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 9640 | 9622 | 9641 | 9695
Participants | 4901 | 5042 | 5087 | 5090
Statistical Analysis 1: Comparison: Control vs High Risk Only vs High Risk Based on Medical Records vs High Risk Based on Algorithm; This analysis compared all groups that were informed they were high risk (High risk only, High risk based on medical records, High risk based on algorithm) to control patients who were not sent a message. Null hypothesis: informing patients they are high risk for flu and flu-related complications does not increase flu vaccination rate; Alternative hypothesis: informing patients they are high risk for flu and flu-related complications increases flu vaccination rate; Test type: Superiority; p = 0.0035, Regression, Logistic
Statistical Analysis 2: Comparison: High Risk Only vs High Risk Based on Medical Records; Null hypothesis: the High risk only and High risk based on medical records messages are equally effective at promoting ﬂu vaccinations; Alternative hypothesis: there is a difference in effectiveness between High risk only and High risk based on medical records. Separate regressions were run to assess pairwise differences between the high-risk arms (analyses 2, 3, and 4). The Holm method was used to test whether each comparison reached significance; Test type: Superiority; p = .613, Regression, Logistic — The p-value reported is uncorrected, but the Holm method was used to determine whether the p-value reached statistical significance
Statistical Analysis 3: Comparison: High Risk Only vs High Risk Based on Algorithm; Null hypothesis: the High risk only and High risk based on algorithm messages are equally effective at promoting ﬂu vaccinations; Alternative hypothesis: there is a difference in effectiveness between High risk only and High risk based on algorithm messages. Separate regressions were run to assess pairwise differences between the high-risk arms (analyses 2, 3, and 4). The Holm method was used to test whether each comparison reached significance; Test type: Superiority; p = 0.889, Regression, Logistic — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: High Risk Based on Medical Records vs High Risk Based on Algorithm; Null hypothesis: the High risk based on medical records and High risk based on algorithm messages are equally effective at promoting ﬂu vaccinations; Alternative hypothesis: there is a difference in effectiveness between High risk based on medical records and High risk based on algorithm messages. Separate regressions were run to assess pairwise differences between the high-risk arms (analyses 2, 3, and 4). The Holm method was used to test whether each comparison reached significance; Test type: Superiority; p = .714, Regression, Logistic — [p-value comment as in outcome 1, analysis 2]

2. Primary Outcome: Flu Vaccination Rate by Risk Level
Description: Patient received a flu vaccination
  Note: For patients who received risk communications, those in the top 3% were always told they were in the top 3% of risk. Those in the top 4-10% of risk were randomized to be told that they were in the top 10% of risk or high risk.
  Control patients in the top 3% and top 4-10% of risk were allocated to the top 3% and randomized to either top 10% or high risk groups, respectively, at the same time as those in the patient contact groups, even though these control patients were not contacted.
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 9640 | 9622 | 9641 | 9695
Participants
  Top 3%: number analyzed (Participants) | 2906 | 2867 | 2855 | 2863
  Top 3% | 1485 | 1536 | 1513 | 1537
  Top 10%: number analyzed (Participants) | 3347 | 3377 | 3389 | 3380
  Top 10% | 1658 | 1749 | 1795 | 1799
  High risk: number analyzed (Participants) | 3387 | 3378 | 3397 | 3452
  High risk | 1758 | 1757 | 1779 | 1754
Statistical Analysis 1: Comparison: High Risk Only vs High Risk Based on Medical Records vs High Risk Based on Algorithm; This analysis tested whether vaccination differed in patients with the same risk level who were sent messages with a vague verbal ("high risk") vs. specific numeric ("top 10%") risk framing. This analysis was limited to those informed they were high risk (High risk only, High risk based on medical records, High risk based on algorithm); Test type: Superiority; p = .181, Regression, Logistic — This p-value is from the same regression as the top 10% risk vs. top 3% risk contrast (analysis 2)
Statistical Analysis 2: Comparison: High Risk Only vs High Risk Based on Medical Records vs High Risk Based on Algorithm; This analysis tested whether vaccination differed in patients with the same numeric risk phrasing are differentially affected due to different specific risk levels (3% vs. 10%). This analysis was limited to those informed they were high risk (High risk only, High risk based on medical records, High risk based on algorithm); Test type: Superiority; p = .301, Regression, Logistic — This p-value is from the same regression as the high risk vs. top 10% risk contrast (analysis 1)

3. Primary Outcome: High Confidence Flu Diagnosis Rate
Description: Patient received a flu diagnosis via a positive PCR/antigen/molecular test
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: Flu cases and other related outcomes (flu complications, ER visits for flu, hospitalizations for flu) in the 2020-2021 flu season were too low to detect any meaningful differences across study arms. Therefore, the study team did not collect data for this outcome.
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: "Likely Flu" Diagnosis Rate
Description: Patient received a diagnosis that was likely flu, as assessed via ICD codes or Tamiflu administration or positive PCR/antigen/molecular test. Note that this outcome is a superset of the "high confidence flu diagnosis rate" outcome.
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: as for outcome 3
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Flu Complications Rate
Description: Patient was diagnosed with flu-related complications
Time Frame: Through 3 months after the end of the flu season (August 31st 2021), approximately 12 months assessment duration
Population: as for outcome 3
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Change in ER Visits From Pre- to Post-intervention
Description: Number of patient visits to the ER, examining relative rate of visits across Time 1 and 2
Time Frame: Within 12 months pre-intervention (Time 1) and within 12 months post-intervention (Time 2)
Population: as for outcome 3
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Change in Hospitalizations From Pre- to Post-intervention
Description: Number of patient hospital visits, examining relative rate of visits across Time 1 and 2
Time Frame: Within 12 months pre-intervention (Time 1) and within 12 months post-intervention (Time 2)
Population: as for outcome 3
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Flu Vaccination Among Fellow Household Members
Description: Non-targeted fellow household members of targeted patients received a flu vaccination
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: Household members were excluded from analysis if they were vaccinated prior to the study start date or if they were contraindicated for flu vaccine. Household members who shared an address with multiple patients in the intervention were counted in this outcome once for every eligible target participant who shared their address.
Measure: Count of Participants; unit: Participants
Groups:
- Control - Household Members: This group had the same address in the EHR as patients in the control group, who received no additional pro-vaccination intervention beyond the health system's normal efforts.
- High Risk Only - Household Members: This group had the same address in the EHR as patients in the high risk only group, who received messages telling them they had been identified to be at high risk for flu complications without specifying how or why the health system believed this to be the case.
- High Risk Based on Medical Records - Household Members: This group had the same address in the EHR as patients in the high risk based on medical records group, who received messages telling them they had been identified to be at high risk for flu complications via analysis of their medical records.
- High Risk Based on Algorithm - Household Members: This group had the same address in the EHR as patients in the High risk based on algorithm group, who received messages telling them they had been identified to be at high risk for flu complications via analysis of their medical records by an AI/ML system.
Arm/Group | Control - Household Members | High Risk Only - Household Members | High Risk Based on Medical Records - Household Members | High Risk Based on Algorithm - Household Members
Number analyzed (Participants) | 7584 | 7981 | 7773 | 7516
Participants | 2136 | 2207 | 2165 | 2175

9. Secondary Outcome: High Confidence Flu Diagnosis Among Fellow Household Members
Description: Non-targeted fellow household members of targeted patients received a flu diagnosis (via a positive PCR/antigen/molecular test)
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: as for outcome 3
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: "Likely Flu" Diagnosis Among Fellow Household Members
Description: Non-targeted fellow household members of targeted patients received a diagnosis that was likely flu (as assessed via ICD codes or Tamiflu administration or positive PCR/antigen/molecular test)
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: as for outcome 3
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Flu Complications Among Fellow Household Members
Description: Non-targeted fellow household members of targeted patients were diagnosed with flu-related complications
Time Frame: Through 3 months after the end of the flu season (August 31st 2021), approximately 12 months assessment duration
Population: as for outcome 3
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Flu Vaccination Among Those at Sub-threshold Risk
Description: Non-targeted sub-threshold risk patients received a flu vaccination
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-threshold Patients
Number analyzed (Participants) | 40030
Participants | 18268

13. Secondary Outcome: High Confidence Flu Diagnosis Among Those at Sub-threshold Risk
Description: Non-targeted sub-threshold risk patients received a flu diagnosis (via a positive PCR/antigen/molecular test)
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: as for outcome 3
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: "Likely Flu" Diagnosis Among Those at Sub-threshold Risk
Description: Non-targeted sub-threshold risk patients received a diagnosis that was likely flu (as assessed via ICD codes or Tamiflu administration or positive PCR/antigen/molecular test)
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: as for outcome 3
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Flu Complications Among Those at Sub-threshold Risk
Description: Non-targeted sub-threshold risk patients were diagnosed with flu-related complications
Time Frame: Through 3 months after the end of the flu season (August 31st 2021), approximately 12 months assessment duration
Population: as for outcome 3
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Post Hoc Outcome: Flu Vaccination Rate by Race
Description: Patient received a flu vaccination
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 9640 | 9622 | 9641 | 9695
Participants
  American Indian or Alaska Native: number analyzed (Participants) | 20 | 20 | 12 | 18
  American Indian or Alaska Native | 6 | 9 | 6 | 7
  Asian: number analyzed (Participants) | 27 | 28 | 23 | 22
  Asian | 19 | 14 | 15 | 13
  Black or African American: number analyzed (Participants) | 336 | 347 | 355 | 372
  Black or African American | 115 | 134 | 143 | 142
  Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 16 | 23 | 16 | 23
  Native Hawaiian or Other Pacific Islander | 5 | 9 | 7 | 7
  White: number analyzed (Participants) | 9233 | 9192 | 9229 | 9249
  White | 4751 | 4871 | 4916 | 4914
  Unknown: number analyzed (Participants) | 8 | 12 | 6 | 11
  Unknown | 5 | 5 | 0 | 7

17. Post Hoc Outcome: Flu Vaccination Rate by Gender
Description: Patient received a flu vaccination
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 9640 | 9622 | 9641 | 9695
Participants
  Female: number analyzed (Participants) | 6278 | 6285 | 6312 | 6266
  Female | 3118 | 3245 | 3235 | 3197
  Male: number analyzed (Participants) | 3362 | 3337 | 3329 | 3429
  Male | 1783 | 1797 | 1852 | 1893

18. Post Hoc Outcome: Flu Vaccination Rate by Ethnicity
Description: Patient received a flu vaccination
Time Frame: Through the the end of the flu season (May 31st 2021), approximately 9 months assessment duration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
Number analyzed (Participants) | 9640 | 9622 | 9641 | 9695
Participants
  Hispanic or Latino: number analyzed (Participants) | 339 | 406 | 354 | 362
  Hispanic or Latino | 118 | 173 | 136 | 146
  Not Hispanic or Latino: number analyzed (Participants) | 9289 | 9196 | 9272 | 9314
  Not Hispanic or Latino | 4778 | 4860 | 4943 | 4938
  Unable to obtain: number analyzed (Participants) | 12 | 20 | 15 | 19
  Unable to obtain | 5 | 9 | 8 | 6

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored. See description.
Description: This is a minimal risk study, and has received expedited IRB review in keeping with 45 CFR §46.110. EHR and claims data will report inputs (i.e., the subject's assigned arm) and outcomes (i.e., flu vaccination, flu diagnosis, flu-like symptoms); we will therefore be unable to monitor this data for AE/SAEs other than the study outcomes themselves.
Arm/Group | Control | High Risk Only | High Risk Based on Medical Records | High Risk Based on Algorithm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
One primary and multiple secondary outcomes involved analysis of flu diagnoses and complications. However, flu cases and other related outcomes in the 2020-2021 flu season were too low to detect any difference in these more distal outcomes, so results are limited to flu vaccination outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT04323137/Prot_001.pdf
  • Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT04323137/SAP_000.pdf